CLINICAL TRIAL: NCT00884481
Title: A Multi-centre and Prospective Trial to Evaluate the Effects on Multiple Sclerosis Related Fatigue During Treatment With Tysabri in Patients With Relapsing Remitting Multiple Sclerosis Over the Course of 12 Months
Brief Title: Effects of Tysabri (BG00002) Over 12 Months on MS Related Fatigue in Participants With RRMS
Acronym: TYNERGY
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: TYNERGY; 2008-008065-35 (EudraCT Number); NCT00966797 (obsolete NCT alias)
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Natalizumab: Participants with MS treated with Tysabri over 12 months
  Interventions: Other: Natalizumab

INTERVENTIONS:
Other: Natalizumab — Participants treated with Tysabri
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of this trial is to observe the Multiple Sclerosis (MS) related fatigue during treatment with Tysabri as measured by changes in the fatigue scale for motor and cognitive functions (FMSC) over the course of 12 months. The secondary objectives are: To investigate changes in fatigue, capacity for work, Health Related Quality of Life (HRQol), sleepiness, cognitive impairment, physically activity induced exhaustion, speed of walking, status of MS disease progression and amount of walking at different times points after initiation of Tysabri treatment in participants diagnosed with Relapsing-Remitting Multiple Sclerosis (RRMS). Changes in fatigue are measured at 3, 6 and 9 months, whereas changes in capacity for work, HRQoL, sleepiness, cognitive impairment, physical activity induced exhaustion, speed of walking, status of MS disease progression and amount of walking are measured at 6 and 12 months. To investigate correlation between fatigue and cognitive impairment, depression and physically activity induced exhaustion and status of MS disease progression in participants at baseline, 6 and 12 month of treatment with Tysabri and to document any changes in fatigue related medication.

ELIGIBILITY:
Key Inclusion Criteria:

* Tysabri prescribed according to national guidelines but not yet started treatment
* Signed informed consent form
* FSMC sum score above > 43 at baseline (mild fatigue)

Key Exclusion Criteria:

* FSMC sum score below 43 at baseline
* History of treatment with Tysabri
* EDSS > 6 at baseline
* Amphetamine as medication
* Major depression

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Relapsing Remitting Multiple Sclerosis initiating treatment with Tysabri
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
To investigate the MS related fatigue during treatment with Tysabri as measured by changes in the fatigue scale for motor and cognitive functions (FMSC) over the course of 12 months. | 0 month and 12 months
  A fatigue scale for motor and cognitive functions (FSMC) has been developed and validated by Penner et al. FSMC differentiates between motor and cognitive fatigue and is less susceptible to confounding by depression. Thus, FSMC is more specific in measuring MS-related fatigue.

SECONDARY OUTCOMES:
Changes in fatigue after initiation of Tysabri treatment | 3 months, 6 months, 9 months
Change in capacity for work (capacity for work questionnaire (CWQ)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  Capacity for Work Questionnaire (CWQ) is used to collect data regarding number of working hours and sickness absence.
Change in health-related-quality of life (HRQ0L) (short form-12 questions (SF-12)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall HRQOL. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Change in Sleepiness (Epworth sleepiness scale (ESS)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The ESS is a self-administered 8-item questionnaire with that provides a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. Each question is rated on a 4-point scale (0 - 3), their usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily lives, although not necessarily every day. The total ESS score is the sum of 8 item-scores and can range between 0 and 24, where higher scores indicate higher levels of a person's level of daytime sleepiness.
Change in cognitive impairment (the paced auditory serial addition test (PASAT) and symbol digit modalities test (SDMT)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The PASAT is the third and last component of the MSFC. SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best).
Change in depression (Center for epidemiologic studies depression scale (CES-D)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  CES-D is a self-report measure of depression severity.
Change in Physical activity induced exhaustion (Borg scale CR10 (BS-CR10)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The Borg Scale measures perceived exertion. It is used to document the patient's exertion during a test. It ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion.
Change in speed of walking (6MWT) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Change in status of MS disease progression (expanded disability status scale (EDSS)) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Change in amount of walking (step counter) at different points after initiation of Tysabri treatment | 0, 6 months, 12 months
To investigate correlation between fatigue and cognitive impairment, depression and physically activity induced exhaustion and status of MS disease progression | 6 months, 12 months
To document any changes in fatigue related medication | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (27):
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Villach
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Odense
- Norway (7):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Drammen
  - Research Site, Førde
  - Research Site, Lillehammer
  - Research Site, Molde
  - Research Site, Oslo
- Sweden (12):
  - Research Site, Danderyd
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Norrköping
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Umeå

REFERENCES:
- [Result] Wickstrom A, Dahle C, Vrethem M, Svenningsson A. Reduced sick leave in multiple sclerosis after one year of natalizumab treatment. A prospective ad hoc analysis of the TYNERGY trial. Mult Scler. 2014 Jul;20(8):1095-101. doi: 10.1177/1352458513517590. Epub 2013 Dec 30. PMID 24378984
- [Result] Svenningsson A, Falk E, Celius EG, Fuchs S, Schreiber K, Berko S, Sun J, Penner IK; Tynergy Trial Investigators. Natalizumab treatment reduces fatigue in multiple sclerosis. Results from the TYNERGY trial; a study in the real life setting. PLoS One. 2013;8(3):e58643. doi: 10.1371/journal.pone.0058643. Epub 2013 Mar 21. PMID 23555589
- [Result] Penner IK, Sivertsdotter EC, Celius EG, Fuchs S, Schreiber K, Berko S, Svenningsson A; TYNERGY trial investigators. Improvement in Fatigue during Natalizumab Treatment is Linked to Improvement in Depression and Day-Time Sleepiness. Front Neurol. 2015 Feb 23;6:18. doi: 10.3389/fneur.2015.00018. eCollection 2015. PMID 25755648